Neuroimaging in Patients Undergoing TMS for Depression

NCT02974296

Document Date: June 17, 2019

Statistics: Pre-planned analyses focused on mixed effect regression models to test whether change in rsfc pre/post both sdTMS and pgTMS differs by treatment group. Association between change in HDRS and that of each rsfc was measured using linear regression. Group difference in the association was tested by adding the interaction term between change in rsfc and treatment group. Fisher's z transform was applied to individual rsfc maps before group level analyses; corrected p-values using FDRs controlled multiple comparison correction were computed (see Suppl. Methods for further details). Bartlett's test was performed to test variance homogeneity across groups. Wherever equal variance hypothesis was rejected, we refit the model allowing different variance by group.